CLINICAL TRIAL: NCT01088737
Title: An Open Monocentric Pilot Study to Investigate the Potential of Imiquimod 5% Cream to Detect Residual and to Prevent Recurrence of Lentigo Maligna After Surgical Excision
Brief Title: Imiquimod to Detect Residual Lesions and Prevent Recurrence of Lentigo Maligna
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Trial Photoderm Graz 2010-1
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Lentigo Maligna
Keywords: Lentigo maligna; melanoma; imiquimod; prevention
MeSH Terms: conditions — Hutchinson's Melanotic Freckle; Melanoma | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imiquimod — Imiquimod 5% cream is applied once daily. Each patient will begin with the application 3x/week. After two weeks of treatment the inflammation response to imiquimod will be assessed. If no or only minor inflammation is detectable in the treatment area, the dosing schedule will be increased to 5x/week. After four weeks of treatment the inflammation response will be assessed again. If still no or only minor inflammation is detectable, application will be extended to daily use.
  Other Names: Aldara

SUMMARY:
This is a prospective, longitudinal, uncontrolled study with follow-up for 5 years.Patients having undergone surgical excision of lentigo maligna (LM) or lentigo maligna melanoma (LMM) will be invited to this study. Eligible patients will start treatment with imiquimod 6 weeks after the excision, the treatment will last for up to 12 weeks. Inflammatory reactions and the occurrence of residual lesions will be documented. The healing effect will be determined (initial clearance rate) 20 weeks after start of treatment with imiquimod. All patients who were enrolled (=exposed to imiquimod in this study) will be followed up for 5 years or until recurrence of the LM or LMM

DETAILED DESCRIPTION:
Imiquimod (Aldara) 5% cream will be applied starting 6 weeks post-surgery to an area within 5 cm of treatment margins to each side of the original scar of the LM or LMM excision. Time period between removal of stitches and first administration of imiquimod should be 4 weeks, correspondent to approximate 6 weeks post surgery. Imiquimod cream is applied once daily. Each patient will begin with the application 3x/week. After two weeks of treatment the inflammation response to imiquimod will be assessed. If no or only minor inflammation is detectable in the treatment area, the dosing schedule will be increased to 5x/week. After four weeks of treatment the inflammation response will be assessed again. If still no or only minor inflammation is detectable, application will be extended to daily use. An interruption of the treatment with imiquimod cream is considered if severe local inflammatory reaction occurs, severe systemic reactions are apparent or if super-infection is observed at the treatment area. The primary objective of the study is to investigate the potential of imiquimod 5% cream to eliminate possible subclinical lesions of LM that resides after surgical excision by determining the long-term recurrence rates. Secondary objectives of the study describe the incidence of subclinical residual lesions and local skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Having undergone surgical excision of LM or LMM
* Positive histological finding of LM or LMM (positive histology of primary excision)

Exclusion Criteria:

* History of allergic reaction to imiquimod or its excipients.
* Pregnancy, breast-feeding or planned pregnancy during the study and women of child-bearing potential not using adequate contraception. Women of child bearing potential not using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, tubal ligation or vasectomised partner
* History of malignant melanoma having metastasised or where metastasis could be expected
* Other malignant tumours in the study treatment area (exception actinic keratosis (AK))
* Lack of ability or willingness to give informed consent
* Lack of willingness to have personal study related data collected, archived or transmitted according to protocol
* Anticipated non-availability for study visits/procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Elimination of possible subclinical lesions of LM that resides after surgical excision by determining the long-term recurrence rates. | 60 months

SECONDARY OUTCOMES:
Incidence of subclinical residual lesions and local skin reactions. | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (2):
- Austria (2):
  - Medical University of Graz, Dept. Dermatology, Graz
  - Medical University of Graz, Graz